CLINICAL TRIAL: NCT06441526
Title: Surgical Closure Versus Anti-TNF in the Treatment of Perianal Fistulas in Crohn's Disease (PISA-II): a Comprehensive Cohort Design
Brief Title: Surgical Closure vs Anti-TNF in the Treatment of Perianal Fistulas in Crohn's Disease (PISA-II): a Comprehensive Cohort Design
Acronym: PISA-II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Willem A. Bemelman, Principal investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL66176.018.18
Record Dates: First submitted 2019-04-10; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Perianal Fistula; Crohn Disease
Keywords: Crohn's disease; Perianal fistula; Anti-TNF; Advancement plasty; LIFT-procedure; Fistula closure; Comprehensive cohort design
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Intervention Model Description: This is an international, multicentre, prospective, comprehensive cohort design trial to identify the most optimal treatment of Crohn's high perianal fistulas. In a comprehensive cohort design patients with a preference will be treated accordingly, whereas only those indifferent to treatment will be randomised in the usual way (combined randomised and preference cohort).
Who Masked: Outcomes Assessor
Masking Description: The primary outcome is fistula closure based on MRI (completely fibrotic fistula tract). A radiologist blinded to treatment allocation will score fibrosis and inflammation of the tract based on MRI.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Anti-TNF (Active Comparator): Seton placement, followed by anti-TNF medication (infliximab or adalimumab) in combination with a immunomodulator after ± 2 weeks. The seton will be removed after ± 6 weeks. Continuation of anti-TNF medication for at least 1 year, after one year continuation is at the discretion of treating physician.
  Interventions: Drug: anti-tumour necrosis factor α antibodies
- Surgical closure (Active Comparator): Seton placement, followed by anti-TNF medication in combination with a immunomodulator after ± 2 weeks. After 8-10 weeks removal of seton and surgical closure (advancement plasty or ligation of the intersphincteric tract (LIFT) procedure). Anti-TNF in combination with a immunomodulator will be stopped after ± 4 months.
  Interventions: Procedure: Advancement plasty

INTERVENTIONS:
Drug: anti-tumour necrosis factor α antibodies — Biological drug
  Arms: Anti-TNF
Procedure: Advancement plasty — Surgical closure of the internal opening
  Other Names: Ligation of the intersphincteric tract (LIFT)
  Arms: Surgical closure

SUMMARY:
Currently, the treatment of Crohn's patients with perianal fistulas predominantly exists of anti-TNF medication. However, its efficiency has never been directly compared to surgical closure of the perianal fistula. The aim of this study is to compare radiological fistula healing at MRI after 18 months follow-up in Crohn's patients undergoing surgical closure to anti-TNF medication as treatment of perianal Crohn's fistulas.

Study design: In this multicenter comprehensive cohort design (CCD) Crohn's patients with a (re)active high perianal fistula will be allocated to anti-TNF for 1 year or surgical closure after 2 months under a short course of anti-TNF. Patients with a distinct preference will be treated accordingly, whereas only indifferent patients will be randomised in the usual way.

Main study parameters/endpoints: The primary outcome parameter is the number of patients with radiologically closed fistulas based on an evaluated MRI-score after 18 months. Secondary outcomes are clinical closure, number of patients undergoing surgical re-interventions and number of re-interventions, recurrences and quality of life based on the Perianal Disease Activity Index (PDAI).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: All patients will receive one of the two standard treatment approaches that are currently used for Crohn's fistulas. All effort has been performed to ensure most optimal treatment, according to best available evidence and current guidelines. Since there is no experimental study-arm, there are no additional risks associated with participation. During the study, the medical staff and trial nurses will monitor the necessity of surgical interventions and hospitalizations. At baseline and after 18 months all patients will undergo a MRI to score the fistula. Secondary outcome parameters will be assessed during visits to the outpatient clinic or telephone consultations at baseline and at intervals of 3 months for the duration of the study period. Every 6 months patients were asked to fill out the PDAI questionnaire with their physician. Based on the available literature, radiological closure of fistulas is expected in 40% of patients in the surgical closure group compared to 15% in the anti-TNF group. The increase in closure rate from 15% to 40% is considered clinically relevant. Due to the combination of a preference and randomized cohort, the appropriate sample size to detect this 25% difference is flexible and is adjusted for a skewed distribution. The minimal sample size, in case of a 1:1 treatment allocation, needed to detect this difference with a Chi-square test equals 86 patients (alpha 0.05, power 80%). The maximal allowed skewed distribution is set at 1:4, which will result in a maximal sample size of 116 patients.

ELIGIBILITY:
Inclusion criteria

* ≥ 18 years
* (re-)active perianal fistula
* High perianal fistula tract (intersphincteric, transsphincteric, suprasphincteric) located in the upper two-thirds of the external sphincter or puborectal muscle
* Fistula with one internal opening (based on MRI imaging). The number of external fistulas does not have to be taken into account
* Written informed consent

4.3 Exclusion criteria

* Proctitis (defined as any active mucosal inflammation or ulcer > 5mm in the rectum)
* Anorectal stenosis (defined as the impossibility to introduce a proctoscope)
* Submucosal fistulas & low intersphincteric fistulas (lower one-third of external sphincter)
* Rectovaginal fistula
* Multiple internal openings
* Use of Anti-TNF medication for more than 3 months
* Previous failure of Anti-TNF treatment for perianal fistula
* Patients with a stoma
* Dementia or altered mental status that would prohibit the understanding and giving of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2013-09-14 (Actual); Primary Completion 2019-12-07 (Actual); Study Completion 2021-06-07 (Actual)

PRIMARY OUTCOMES:
Fistula closure | at 1,5 year
  The number of patients with radiologically closed (completely fibrotic) fistula tract on MRI

SECONDARY OUTCOMES:
Clinical closure | at 1,5 year
  The number of patients with clinical closure, defined as closure of the external opening without discharge of pus or faeces on palpation
The number of patients undergoing surgical re-intervention | at 1,5 year
  Amount of patients undergoing surgical re-intervention
The number of re-intervention | at 1,5 year
  Amount of re-interventions
The quality of life of a patient | Every six months from baseline till 18 months
  measured by the Perianal Disease Activity Index (PDAI score)
The number of recurrences | at 1,5 year
  Amount of patients with a recurrence, defined as re-opening of the external opening after clinical closure

CONTACTS AND LOCATIONS:
Overall Officials: Willem Bemelman, MD PhD, Principal Investigator — Amsterdam UMC, location AMC
Locations (1):
- Amsterdam UMC, Amsterdam-Zuidoost, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol